CLINICAL TRIAL: NCT04261049
Title: Effect of ZILRETTA Injection on Neuromuscular Function, Gait Biomechanics and Physical Performance
Brief Title: Effect of Zilretta Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19-3562
Record Dates: First submitted 2020-02-05; First posted 2020-02-07 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2020-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZILRETTA Injection (Experimental): All patients upon enrolling in the study will receive a single 5 mL injection of 32 mg ZILRETTA into the affected knee joint.
  Interventions: Drug: Triamcinolone Acetonide Extended-Release Injectable Suspension

INTERVENTIONS:
Drug: Triamcinolone Acetonide Extended-Release Injectable Suspension — A single ZILRETTA® (triamcinolone acetonide extended-release injectable suspension) intra-articular knee injection.
  Other Names: Zilretta Injectable Product

SUMMARY:
The purpose of this study is to examine the pre-post effects of a single ZILRETTA knee injection on physiological measures of self-reported pain and disability, physical performance, and physical activity in individuals with knee osteoarthritis (OA). The investigators will recruit 35 symptomatic knee OA patients for this study. All data will be collected prior to injection (baseline), as well as at 4 (post 1) and 8-week follow-ups (post 2).

DETAILED DESCRIPTION:
Individuals with knee osteoarthritis (OA) demonstrate significant physical disability which leads to diminished physical activity, a lesser quality of life, as well as a higher risk of inactivity related comorbidities including mortality. This is thought to be caused by an inability to voluntarily activate your quadriceps muscle due, in part, to knee joint swelling and joint-related pain. Incomplete muscle activation causes quadriceps weakness.

Individuals with quadriceps weakness exhibit changes in their walking biomechanics which is associated with diminished physical function and lesser physical activity in those with knee OA. Therefore, it is critical to develop interventions that target mechanisms causing decreased quadriceps activation in order to restore optimal walking biomechanics and improve physical activity.

The ZILRETTA knee injection is an FDA approved, extended release corticosteroid for in patients with knee osteoarthritis and has been shown to reduced knee pain for 3 months in approximately 70% of patients. Currently, there are no studies that have examined ZILRETTA's objective effectiveness on physical activity, biomechanics, and performance tests in patients who have received an injection.

The overall purpose of the current study is to examine the effect of a ZILRETTA knee injection on functional and performance tests including quadriceps neuromuscular activation, quadriceps strength, walking gait biomechanics, and a battery of physical performance outcomes at 4 and 8-weeks following injection in 35 individuals with knee OA.

ELIGIBILITY:
Full Inclusion Criteria:

* Male or female between the ages of 40 and 75 years old who:
* Exhibit symptomatic knee OA, defined as a normalized WOMAC function subscale score >31(out of 100 points, indicating highest degree of dysfunction)
* Have radiographic evidence of tibiofemoral OA (2-4 on the Kellgren-Lawrence scale)
* Provide written informed consent and the ability to comply with the requirements of the study.
* Be willing to abstain from use of the following protocol-restricted medications during the study:

  * Corticosteroid injections into the knee or any lower extremity joint will be restricted for 3 months prior to the screening visit (based on the drug half-life) and throughout the entirety of the study period including the 8-week follow-up test. Information about when the latest corticosteroid injection occurred for each participant prior to screening in order to determine when each participant can attend the screening visit.
  * Hyaluronic acid injections into the knee or any lower extremity joint will be restricted for 6 months prior to the screening visit (based on the drug half-life) and throughout the entirety of the study period including the 8-week follow-up test. Information about when the latest hyaluronic acid injection occurred for each participant prior to screening in order to determine when each participant can attend the screening visit.
  * Prescription Depressants (Examples: opiates and opioids, barbiturates, tranquilizers and benzodiazepines) will be restricted 4-weeks prior to screening and throughout the study period as these medications may affect the neuromuscular function.
  * Prescription Stimulants (Example: amphetamines) will be restricted 4-weeks prior to screening and throughout the study period as these medications may affect the neuromuscular function
  * Non-steroidal anti-inflammatory drugs (NSAIDs) will be restricted 24 hours prior to screening or follow-up testing sessions. NSAID use will be tracked and patients instructed not to change their NSAIDs usage during the 8-weeks of the study.
  * Acetaminophen will be restricted 24 hours prior to screening or follow-up testing sessions. Acetaminophen use will be tracked and patients instructed not to change their Acetaminophen usage during the 8-weeks of the study.

Full Exclusion Criteria:

Potential participants meeting any of the following criteria (based on the electronic medical record or in laboratory screening) will be excluded if they:

* Are hypersensitive to triamcinolone acetonide, corticosteroids or any components of the product
* Have other intra-articular investigational drug/biologic use in the previous 6-months
* Have been diagnosed with a cardiovascular condition restricting exercise
* Have had a corticosteroid injection in the involved knee in the previous 3-months or hyaluronic acid injection in the involved knee in the previous 6-months
* Have a pacemaker
* Have a neurodegenerative condition
* Have rheumatoid arthritis
* Have diabetes
* Have cancer
* Have a neural sensory dysfunction over the knee
* Have a body mass index (BMI) over 35
* Have a history of lower extremity orthopaedic surgery in the past year
* Have a history of a traumatic knee injury in the past 6 months
* Have any history of total knee arthroplasty in either extremity
* Have a diagnosed, non-reconstructed knee ligament tear
* Need an assistive device to walk
* Are currently pregnant or planning to become pregnant while enrolled in the study
* Are taking medications that can react harmfully with injected corticosteroids

NOTE: Individuals that have bilateral knee OA will not be excluded unless they meet another exclusion criteria. In case a patient needs an injection in both knees, they will be excluded. Only one knee will be injected for this study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Percentage Change in Mean Maximal Quadriceps Strength as Measured by the Maximal Isometric Voluntary Contractions Normalized to Body Weight from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  Quadriceps strength was measured in Newton Meters normalized to body weight of the individuals. Strength was assessed in 90 degrees of knee flexion.
Percentage Change in Mean Voluntary Quadriceps Activation as Measured by the Central Activation Ratio Expressed as a Percent of Full Activation from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  The investigators assessed voluntary quadriceps central activation ratio as a representative variable of lower extremity neuromuscular activation using the supra imposition technique. Quadriceps central activation ratio has been demonstrated to be significantly decreased in knee osteoarthritis (OA) compared to healthy, matched controls, and the investigators have reported acceptable measurement reliability (ICC2,k = 0.85)
Percentage Change in Mean Knee Flexion Angle During Walking Gait Measured in Degrees of Knee Flexion from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  The peak Knee Flexion Angle was calculated using using inverse dynamics calculations in the first 50% of the stance phase of gait and during self selected gait speed.
Percentage Change in Mean Internal Knee Extension Moment During Walking Gait Measured in Nm/ Body Weight*m from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  The peak internal knee extension moment was calculated using using inverse dynamics calculations in the first 50% of the stance phase of gait and normalized to the Body Weight* height (m) of the individual during self selected gait speed.
Percentage Change in Mean of Self-reported Disability Score as Measured by the Western Ontario and McMasters Universities Index from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  The Western Ontario and McMasters Universities Index is reliable and valid measure of self reported disability. The physical function consists of 17 items and asks about the magnitude of difficulty when ascending and descending stairs, rising from sitting, standing, bending, walking, getting in / out of a car, shopping, putting on and taking off socks, rising from bed, lying in bed, getting in and out of the bath, sitting, getting on and off the toilet, completing heavy household duties, and completing light household duties. Each item is presented in a 5 point Likert-type format and uses the following descriptors for possible answer choices none, mild moderate, severe, and extreme. Each descriptor corresponds to an ordinal scale of 0-4. The scores are summed for the items in each subscale, with total possible ranges as 0-68. Higher scores on the WOMAC indicate greater amounts of functional limitations.
Percentage Change in mean of self-reported Disability Score as Measured by the Knee Injury and Osteoarthritis Outcome Score from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  The Knee Injury and Osteoarthritis Outcomes Score (KOOS) consists of five subscales: Pain (9 items), Symptoms (7 items), Function in Activities of Daily Living (17 items), Function in Sport and Recreation (5 items) and Knee Related Quality of Life (4 items). Each item is presented in a 5 point Likert-type format that ranges from 0 (no problems) to 4 (extreme problems). Totals from each subscale are transformed to a 0-100 score. Lower scores on the KOOS indicate greater amounts of functional limitations.
Percentage Change in Physical Activity Scale for the Elderly from baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  Physical Activity Scale for the Elderly (PASE) scores are calculated from weights and frequency values for each of 12 types of activity. Responses to the first question about sitting activities are not scored. The scale is continuous with higher scores indicating greater physical activity.
Percentage Change in 30-s chair-stand test from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  The number of times that an individual can sit and stand in 30 seconds.
Percentage Change in 20 meter fast-paced walk test from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  The investigators will time the amount of seconds it takes to walk 20 meters.
Percentage Change in Stair-climb test from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  The investigators will time the amount of seconds it takes to walk up and down a flight of stairs.
The percentage change in steps per day from Baseline to the 8-week follow-up. | Baseline and 8-week follow-up
  Physical activity will be measured in the form of steps per day using an ActiGraph accelerometer. Participants will wear the ActiGraph for 7 days following each testing session.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pietrosimone, PhD, ATC, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- MOTION Science Institute, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Elliott P, Hawthorne G. Imputing missing repeated measures data: how should we proceed? Aust N Z J Psychiatry. 2005 Jul;39(7):575-82. doi: 10.1080/j.1440-1614.2005.01629.x. PMID 15996138
- [Background] Harkey MS, Gribble PA, Pietrosimone BG. Disinhibitory interventions and voluntary quadriceps activation: a systematic review. J Athl Train. 2014 May-Jun;49(3):411-21. doi: 10.4085/1062-6050-49.1.04. Epub 2014 Feb 3. PMID 24490843
- [Background] Hopkins JT, Ingersoll CD, Edwards JE, Cordova ML. Changes in soleus motoneuron pool excitability after artificial knee joint effusion. Arch Phys Med Rehabil. 2000 Sep;81(9):1199-203. doi: 10.1053/apmr.2000.6298. PMID 10987162
- [Background] Hopkins J, Ingersoll CD, Edwards J, Klootwyk TE. Cryotherapy and Transcutaneous Electric Neuromuscular Stimulation Decrease Arthrogenic Muscle Inhibition of the Vastus Medialis After Knee Joint Effusion. J Athl Train. 2002 Mar;37(1):25-31. PMID 12937440
- [Background] Hopkins JT, Ingersoll CD, Krause BA, Edwards JE, Cordova ML. Effect of knee joint effusion on quadriceps and soleus motoneuron pool excitability. Med Sci Sports Exerc. 2001 Jan;33(1):123-6. doi: 10.1097/00005768-200101000-00019. PMID 11194097
- [Background] Jones CJ, Rikli RE, Beam WC. A 30-s chair-stand test as a measure of lower body strength in community-residing older adults. Res Q Exerc Sport. 1999 Jun;70(2):113-9. doi: 10.1080/02701367.1999.10608028. PMID 10380242
- [Background] KELLGREN JH, LAWRENCE JS. Radiological assessment of osteo-arthrosis. Ann Rheum Dis. 1957 Dec;16(4):494-502. doi: 10.1136/ard.16.4.494. No abstract available. PMID 13498604
- [Background] Kennedy DM, Stratford PW, Wessel J, Gollish JD, Penney D. Assessing stability and change of four performance measures: a longitudinal study evaluating outcome following total hip and knee arthroplasty. BMC Musculoskelet Disord. 2005 Jan 28;6:3. doi: 10.1186/1471-2474-6-3. PMID 15679884
- [Background] Lewek M, Rudolph K, Axe M, Snyder-Mackler L. The effect of insufficient quadriceps strength on gait after anterior cruciate ligament reconstruction. Clin Biomech (Bristol). 2002 Jan;17(1):56-63. doi: 10.1016/s0268-0033(01)00097-3. PMID 11779647
- [Background] Leyland KM, Gates LS, Sanchez-Santos MT, Prieto Alhambra D, Judge A, Collins G, Cleveland R, Felson D, Jordon JM, Callahan LF, Nevitt M, Saberi Hosnijeh F, van Meurs JB, Jones G, Newton J, Batt M, Altman D, Cooper C, Arden N, Committee PC. Knee osteoarthritis and the risk of premature mortality in the community: an international individual patient level meta-analysis in 9889 subjects. Osteoarthritis and Cartilage. 2017;25:S29-S30.
- [Background] Liikavainio T, Isolehto J, Helminen HJ, Perttunen J, Lepola V, Kiviranta I, Arokoski JP, Komi PV. Loading and gait symmetry during level and stair walking in asymptomatic subjects with knee osteoarthritis: importance of quadriceps femoris in reducing impact force during heel strike? Knee. 2007 Jun;14(3):231-8. doi: 10.1016/j.knee.2007.03.001. Epub 2007 Apr 23. PMID 17451958
- [Background] Liikavainio T, Lyytinen T, Tyrvainen E, Sipila S, Arokoski JP. Physical function and properties of quadriceps femoris muscle in men with knee osteoarthritis. Arch Phys Med Rehabil. 2008 Nov;89(11):2185-94. doi: 10.1016/j.apmr.2008.04.012. PMID 18996249
- [Background] Luc BA, Lepley AS, Tevald MA, Gribble PA, White DB, Pietrosimone BG. Reliability of corticomotor excitability in leg and thigh musculature at 14 and 28 days. J Sport Rehabil. 2014 Nov;23(4):330-8. doi: 10.1123/jsr.2013-0069. Epub 2013 Oct 1. PMID 24084315
- [Background] Luc BA, Harkey MH, Arguelles GD, Blackburn JT, Ryan ED, Pietrosimone B. Measuring voluntary quadriceps activation: Effect of visual feedback and stimulus delivery. J Electromyogr Kinesiol. 2016 Feb;26:73-81. doi: 10.1016/j.jelekin.2015.10.006. Epub 2015 Nov 2. PMID 26597088
- [Background] Luc-Harkey BA, Blackburn JT, Ryan ED, Harkey MS, Davis HC, Gaynor BR, Nissman DB, Spang JT, Pietrosimone B. Quadriceps Rate of Torque Development and Disability in Persons With Tibiofemoral Osteoarthritis. J Orthop Sports Phys Ther. 2018 Sep;48(9):694-703. doi: 10.2519/jospt.2018.7898. Epub 2018 May 22. PMID 29787693
- [Background] Marcus BH, Selby VC, Niaura RS, Rossi JS. Self-efficacy and the stages of exercise behavior change. Res Q Exerc Sport. 1992 Mar;63(1):60-6. doi: 10.1080/02701367.1992.10607557. PMID 1574662
- [Background] Nuesch E, Dieppe P, Reichenbach S, Williams S, Iff S, Juni P. All cause and disease specific mortality in patients with knee or hip osteoarthritis: population based cohort study. BMJ. 2011 Mar 8;342:d1165. doi: 10.1136/bmj.d1165. PMID 21385807
- [Background] Palmieri-Smith RM, Thomas AC. A neuromuscular mechanism of posttraumatic osteoarthritis associated with ACL injury. Exerc Sport Sci Rev. 2009 Jul;37(3):147-53. doi: 10.1097/JES.0b013e3181aa6669. PMID 19550206
- [Background] Pietrosimone B, Lepley AS, Murray AM, Thomas AC, Bahhur NO, Schwartz TA. Changes in voluntary quadriceps activation predict changes in muscle strength and gait biomechanics following knee joint effusion. Clin Biomech (Bristol). 2014 Sep;29(8):923-9. doi: 10.1016/j.clinbiomech.2014.06.014. Epub 2014 Jul 4. PMID 25062605
- [Background] Pietrosimone BG, McLeod MM, Lepley AS. A theoretical framework for understanding neuromuscular response to lower extremity joint injury. Sports Health. 2012 Jan;4(1):31-5. doi: 10.1177/1941738111428251. PMID 23016066
- [Background] Pietrosimone B, Thomas AC, Saliba SA, Ingersoll CD. Association between quadriceps strength and self-reported physical activity in people with knee osteoarthritis. Int J Sports Phys Ther. 2014 May;9(3):320-8. PMID 24944850
- [Background] Pietrosimone BG, Hertel J, Ingersoll CD, Hart JM, Saliba SA. Voluntary quadriceps activation deficits in patients with tibiofemoral osteoarthritis: a meta-analysis. PM R. 2011 Feb;3(2):153-62; quiz 162. doi: 10.1016/j.pmrj.2010.07.485. PMID 21333954
- [Background] Pietrosimone BG, Saliba SA. Changes in voluntary quadriceps activation predict changes in quadriceps strength after therapeutic exercise in patients with knee osteoarthritis. Knee. 2012 Dec;19(6):939-43. doi: 10.1016/j.knee.2012.03.002. Epub 2012 Apr 13. PMID 22503429
- [Background] Pietrosimone BG, Saliba SA, Hart JM, Hertel J, Kerrigan DC, Ingersoll CD. Effects of disinhibitory transcutaneous electrical nerve stimulation and therapeutic exercise on sagittal plane peak knee kinematics and kinetics in people with knee osteoarthritis during gait: a randomized controlled trial. Clin Rehabil. 2010 Dec;24(12):1091-101. doi: 10.1177/0269215510375903. Epub 2010 Aug 16. PMID 20713439
- [Background] Roos EM, Klassbo M, Lohmander LS. WOMAC osteoarthritis index. Reliability, validity, and responsiveness in patients with arthroscopically assessed osteoarthritis. Western Ontario and MacMaster Universities. Scand J Rheumatol. 1999;28(4):210-5. doi: 10.1080/03009749950155562. PMID 10503556
- [Background] Seeley MK, Park J, King D, Hopkins JT. A novel experimental knee-pain model affects perceived pain and movement biomechanics. J Athl Train. 2013 May-Jun;48(3):337-45. doi: 10.4085/1062-6050-48.2.02. Epub 2013 Feb 20. PMID 23675793
- [Background] Simonsick EM, Gardner AW, Poehlman ET. Assessment of physical function and exercise tolerance in older adults: reproducibility and comparability of five measures. Aging (Milano). 2000 Aug;12(4):274-80. doi: 10.1007/BF03339847. PMID 11073346
- [Background] Tubach F, Ravaud P, Baron G, Falissard B, Logeart I, Bellamy N, Bombardier C, Felson D, Hochberg M, van der Heijde D, Dougados M. Evaluation of clinically relevant states in patient reported outcomes in knee and hip osteoarthritis: the patient acceptable symptom state. Ann Rheum Dis. 2005 Jan;64(1):34-7. doi: 10.1136/ard.2004.023028. Epub 2004 May 6. PMID 15130902
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031